CLINICAL TRIAL: NCT00035542
Title: A Research Study to Determine the Safety and Efficacy of Glucovance Compared to Metformin and Glyburide in Children and Adolescents With Type 2 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Purpose: Treatment
Other Study IDs: CV138-059
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Glucovance; Metformin; Glyburide

INTERVENTIONS:
Drug: Glucovance (metformin HCl/glyburide)
Drug: metformin HCl
Drug: glyburide

SUMMARY:
The purpose of this clinical research study is to see if Glucovance, a medication currently approved for use in adults with type 2 diabetes, can control type 2 diabetes safely and effectively in children 9 to 16 years of age.

ELIGIBILITY:
Children ages 9-16 years with a diagnosis of type 2 diabetes mellitus who are not adequately controlled with diet and exercise, with or without oral hypoglycemic therapy, and have an HbA1c greater than 6.4%

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-12; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (50):
- United States (50):
  - Childrens's Health System/Dept of PED/Diabetes/Endoncrinology, Birmingham, Alabama
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Hazan, Lydie, Beverly Hills, California
  - Bautista Research & Medical Center, Fresno, California
  - Health Care Link, Inc, La Jolla, California
  - Neufeld Medical Group, Los Angeles, California
  - National Institute Of Clinical Research, Los Angeles, California
  - Pasadena Pediatric Endocrinology Diabetes, Pasadena, California
  - A.R.I. Clinical Trials, Redondo Beach, California
  - Sutter Institute For Medical Research, Sacramento, California
  - Children's Hospital, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - EDU Practice Pediatric Endocrinology, Tallahassee, Florida
  - Southeastern Endocrine and Diabetes, Atlanta, Georgia
  - University of Hawaii/Diabetes Research Group, ‘Ewa Beach, Hawaii
  - St. James Diabetes Center, Chicago Heights, Illinois
  - Lutheran General Children's Hospital, Park Ridge, Illinois
  - Raymond Blank Children's Hospital, Des Moines, Iowa
  - Louisville Metabolic & Athersclerosis Research Center/Advanced Cardiovascular Institute, Louisville, Kentucky
  - Bay East Endocrinologists, Easton, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - JM Clinical Trials Inc, Swansea, Massachusetts
  - Center for Health Management, Gulfport, Mississippi
  - Medex Healthcare Research, St Louis, Missouri
  - Diabetes, Endocrine & Nutrition Core Physicians, Hampton, New Hampshire
  - Hackensack Medical Center, Hackensack, New Jersey
  - Endocrine & Diabetes Center, Jersey City, New Jersey
  - SUNY Downstate Medical Center / Dept of Endocrinology, Brooklyn, New York
  - Children's Hospital of Buffalo/Kaledia Health Diabetes Center, Buffalo, New York
  - Winthrop University Hospital, Clinical Trials Center, Mineola, New York
  - St Luke's Roosevelt Hospital/Westside Pediatrics Assoc/Clinical Pharmacology Program, New York, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester/Dpt Pediatrics, S.M.H., Rochester, New York
  - Montefioe Medical Center - DIV / c/o BRANY, The Bronx, New York
  - East Carolina University School of Medicine Dept of Pediatrics, Greenville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Children's Hospital/Dept of Pediatrics, Cleveland, Ohio
  - Forum Health/Western Reserve/TOD Children's Hospital, Youngstown, Ohio
  - Greenville Hospital System/Mountain View Clinical Research/Div of Pediatric Endocrinology, Greenville, South Carolina
  - Lebonheur Children's Medical Center, Memphis, Tennessee
  - South Texas Applied Research, Corpus Christi, Texas
  - Driscoll Children's Hospital/Division of Medical Education/William Riley, Corpus Christi, Texas
  - Tri Quest Research Inc, Houston, Texas
  - Wilford Hall USAF Medical Center, Lackland Air Force Base, Texas
  - Lance Sloan, MD, Lufkin, Texas
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas
  - S.A.M. Clinical Research Center, San Antonio, Texas
  - Monarch Research Associates, Norfolk, Virginia